CLINICAL TRIAL: NCT00236275
Title: PET and MRI in the Follow-up of Neoadjuvant Chemotherapy of Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Pierre and Marie Curie University (Other)
Responsible Party: Zakia IDIR, Department Clinical Research of developpement
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P020907
Record Dates: First submitted 2005-10-11; First posted 2005-10-12 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2007-03

CONDITIONS: Breast Cancer
Keywords: Comparison of imaging modalities; predict the effectiveness of neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Fluoro-L-thymidine-(18F)
  Interventions: Drug: Fluoro-L-thymidine-(18F)

INTERVENTIONS:
Drug: Fluoro-L-thymidine-(18F) — Fluoro-L-thymidine-(18F)

SUMMARY:
Predict and follow thanks to imaging the response to neoadjuvant chemotherapy in locally advanced breast carcinoma. Hypothesis : FLT-(18F)PET will be a predictor superior to both FDG-(18F) PET and MRI

DETAILED DESCRIPTION:
PET/CT with FDG-(18F) and FLT-(18F) and MRI are performed at the initial staging, 3 times during sequential adjuvant chemotherapy and prior to surgery, aiming to find the most efficient modality to predict the response to neoadjuvant chemotherapy of the primary breast cancer and its possible lymph node metastases. Post-surgical histology and a 6 month follow-up (to detect occult metastases) will constitute the standard of truth for determination and comparison of diagnostic performances.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer scheduled for neoadjuvant chemotherapy followed by surgery

Exclusion criteria:

* Indicated chemotherapy without that a curative tumorectomies is foreseen(planned)
* Patient presenting an evolutionary infectious or inflammatory pathology, including an inflammatory breast cancer, being able to be source(spring) of false-positive results(profits) in TEP-FDG
* Patient in the course of radiotherapy or of chemotherapy or operated at the level of the thorax in 4 weeks preceding the date foreseen(planned) by the examination TEP (pose(installation) of implantable room(chamber) excludes)
* Diabetic waits
* Patient already includes in the other protocols of search(research) for Nuclear Medicine or for imaging using ionization radiations
* Patient not having given her lit(enlightened) assent
* Wait among which the surveillance TEP or the MRI during the chemotherapy will be impossible (that is by geographical or professional imperative, or if contraindication in the MRI, ex: port(bearing) of a pacemaker, cochlear magnetic implants, metal foreign bodies cf protocol)
* Of less than 18 years old or pregnant patient.
* Breast cancer stage(stadium) IV
* Biopsy on the already realized mammary tumor, for the period(delay) lower than 15 j.
* In case of alcoholic poisoning or of antecedents of reaction to the injection of ethanol: not inclusion to be discussed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Determine and compare sensitivity and specificity of 3 different modalities for the prediction of effectiveness of neoadjuvant chemotherapy | during de study
  Determine and compare sensitivity and specificity of 3 different modalities for the prediction of effectiveness of neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Noël TALBOT, Pr,MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital TENON, Paris, France